CLINICAL TRIAL: NCT01649882
Title: Ultrasound Evaluation of Endotracheal Tube Depth for Proper Tube Placement in Different Patient Groups
Brief Title: Ultrasound Evaluation of Endotracheal Tube Depth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai Schoenhage (Other)
Responsible Party: Sponsor-Investigator, Kai Schoenhage, Assistant Professor, Anesthesiology Director of Perioperative Services, Director of Liver Transplant Anesthesia, Department of Anesthesiology, University of Arizona
Organization: University of Arizona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0411
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Intubation, Intratracheal
Keywords: endotracheal tube position; intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- US ETT (ultrasound endotracheal tube) (Experimental): Subjects will have a brief (< 15 minutes) ultrasound exam of the neck after intubation. The cuff of the endotracheal tube as well as the aortic arch will be identified. The distance between the two structures will be measured and recorded.
  Interventions: Procedure: US ETT (ultrasound endotracheal tube)

INTERVENTIONS:
Procedure: US ETT (ultrasound endotracheal tube) — Subjects will have a brief (< 15 minutes) ultrasound exam of the neck after intubation. The cuff of the endotracheal tube as well as the aortic arch will be identified. The distance between the two structures will be measured and recorded.
  Other Names: Ultrasound exam

SUMMARY:
Correct positioning of the endotracheal tube (ETT) is crucial to ensure safe ventilation. To date, no test that can verify this right after intubation at the bedside exists. Indirect tests have false negative and positive results leading to complications or at least difficulties in performing effective ventilation of patients.

Bedside ultrasound could fill this need. Although bedside ultrasound may not be possible or useful in routine intubations, it may prove useful in difficult or questionable cases, where current clinical exams/techniques may not offer a reliable indication of endotracheal tube depth.

DETAILED DESCRIPTION:
Ultrasound is able to visualize some parts of the trachea and the ETT therein and although the actual structures of interest (ETT tip and carina) are difficult or impossible to visualize reliably (due to their air contents reflecting ultrasound beams) one can use surrogates:

The cuff of the ETT can be visualized as it is in- or deflated or it can be filled with an air-fluid(saline) mixture to delineate it inside the trachea.

For the same reason (air reflecting ultrasound beams) the carina is difficult to visualize and one can use the aortic arch which is positioned just anterior to it instead.

This study apart from determining feasibility of the method may produce enough data from ultrasound exams to develop/derive a more pre-cise algorithm than available today aiding in positioning the endotracheal tube in regards to anatomic-al landmarks (teeth, gums, lips) even without the use of ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* requiring anesthesia with an endotracheal tube placed for surgical or procedural purposes
* elective or stable and awake for urgent or emergent surgeries

Exclusion Criteria:

* known tracheal deformities
* thoracic aortic aneurysm
* neck/chest tissue thickness making U/S scanning difficult
* severe trauma, head injuries or any procedures that require immediate surgery

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
concomitant visualization of endotracheal tube cuff and aortic arch by ultrasound in situ | 15 minutes

SECONDARY OUTCOMES:
distance between endotracheal tube cuff and aortic arch by ultrasound in situ | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kai Schoenhage, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States